CLINICAL TRIAL: NCT07331545
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single and Multiple Ascending Doses of QL2401 in Healthy Chinese Adult Participants
Brief Title: Safety, Tolerability, PK, PD, and Immunogenicity of QL2401 in Healthy Chinese Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL2401-101
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Dysfunction-Associated Steatohepatitis(MASH)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2401 (Experimental)
  Interventions: Drug: QL2401
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QL2401 — QL2401 is a recombinant fusion protein administered via subcutaneous injection. Participants will receive single or multiple ascending doses of QL2401.
  Arms: QL2401
Drug: Placebo — Matching placebo administered via subcutaneous injection.
  Arms: Placebo

SUMMARY:
This is a first-in-human, Phase I, randomized, double-blind, placebo-controlled clinical trial to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of QL2401 following single and multiple ascending subcutaneous doses in healthy Chinese adults. The study consists of two parts: single ascending dose (SAD) and multiple ascending dose (MAD). Participants will be randomly assigned to receive either QL2401 or placebo. The primary objective is to assess safety and tolerability. Secondary objectives include evaluation of PK parameters in SAD & MAD; exploratory objectives include assessment of PD biomarkers and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants, aged 18 to 45 years at the time of screening.
2. Body weight of males should be ≥50.0kg and body weight of females should be≥45.0kg, BMI 18.5-32.5 kg/m² (Including boundary values)at the time of screening.
3. During the screening and baseline periods, participants with normal laboratory tests, vital sign measurements, physical examination results, 12-lead electrocardiogram, and abdominal B-ultrasound results, or those with abnormalities judged by the investigators as having no clinical significance (MAD section: those with clinically significant lipid indicators and abdominal B-ultrasound results but meeting the following criteria can be included: TC< 7.2mmol/L, LDL-C< 4.9mmol/L, TG< 4.52mmol/L; Abdominal B-ultrasound indicates mild or moderate fatty liver).
4. Participants voluntarily signed the informed consent form before the trial.
5. Willing to use contraception and comply with study procedures.

Exclusion Criteria:

1. Serious, progressive, and uncontrolled diseases, including but not limited to the cardiovascular system, endocrine and metabolic system, immune system, urinary system, digestive system, respiratory system, blood system, gynecological system, nervous system, mental system, and musculoskeletal system, and the researcher determines that the participant is not suitable for this trial;
2. Serious or chronic recurrent gastrointestinal diseases (such as chronic diarrhea, active ulcer, reflux esophagitis), or screening before 12 weeks underwent gastrointestinal surgery;
3. History of acute or chronic pancreatitis, history of symptomatic gallbladder, pancreas injury can lead to high risk factors of acute pancreatitis, or screening blood amylase > 1.5 x upper limit of normal range (ULN);
4. Type 1 diabetes, type 2 diabetes or other types of diabetes;
5. Abnormal liver, renal, or cardiac function
6. Positive for hepatitis B, C, HIV, or syphilis
7. Pregnant or breastfeeding women
8. History of drug or alcohol abuse
9. Use of prescription drugs within 2 weeks prior to dosing
10. According to the researcher's judgment, it may increase the risks related to the research, may interfere with the interpretation of the research results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | From baseline up to 29 days after last dose (SAD) or 57 days after last dose(MAD)
  Safety and tolerability as assessed by the incidence and severity.